CLINICAL TRIAL: NCT03139058
Title: Prevalence of Liver Fibrosis and Cirrhosis in Patients With Squamous Cell Carcinoma of the Head and Neck
Acronym: fibr'HOM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2016_843_0034
Record Dates: First submitted 2017-04-27; First posted 2017-05-03 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Liver Fibroses; Liver Cirrhoses; Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Liver Cirrhosis; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- prevalence of cirrhosis (Other): Study the prevalence of cirrhosis in patients with VADS cancer
  Interventions: Other: Evaluation of the hepatic fibrosis

INTERVENTIONS:
Other: Evaluation of the hepatic fibrosis — Evaluation of the hepatic fibrosis stage by a hepatological assessment (Clinical, biological and imaging)

SUMMARY:
Tobacco and alcohol are the two major risk factors for upper respiratory tract cancer (VADS).

DETAILED DESCRIPTION:
Tobacco and alcohol are the two major risk factors for upper respiratory tract cancer (VADS). Among patients with VADS cancer, more than 60% reported daily alcohol consumption of more than 20 g / d. Such poisoning can be harmful, causing histological lesions of alcoholic liver disease, such as steatosis, alcoholic hepatitis, liver fibrosis and cirrhosis. In a population consuming more than 50 g of alcohol per day for 5 years, the prevalence of severe hepatic fibrosis is between 30% and 40%. In the therapeutic management of a cancer of VADS, the presence of cirrhosis is a prognostic element, increasing the postoperative risk of haemorrhage, surgical site infection and acute renal failure. The search for cirrhosis in the pre-therapeutic assessment is therefore important. The diagnosis of cirrhosis is not a problem when clinical, biological, radiological or endoscopic signs of hepatic insufficiency or portal hypertension are present. Asymptomatic cirrhosis is more difficult to diagnose without liver biopsy. Noninvasive hepatic exploration techniques have recently been developed and validated for the evaluation of liver fibrosis in the context of alcoholic liver disease. Fibroscan® (Echosens, Paris, France) is an imaging device for measuring the liver hardness (hepatic elasticity expressed in kPa), with a strong correlation with the presence of histological fibrosis of the liver. At the threshold of 19.5 kPa, Fibroscan can be used to diagnose cirrhosis with good diagnostic performance (Se 80%, Sp 90%, VPP 93%, VPN 70%) and good inter- and intra-observer reproducibility. Elastometry is a simple, reliable and non-invasive tool to systematically evaluate hepatic fibrosis in patients with VADS cancer. The examination can be performed during a routine care consultation. The post-therapeutic morbidity induced by cirrhosis in the cancers of VADS is not well known and there is no recommendation in France about the hepatic explorations to be carried out during the initial assessment of these neoplasias. It is essential to be able to specify this morbidity in order to adapt if necessary the therapeutic strategy of cancers of VADS.

The objective of this study is to systematically determine the presence of cirrhosis and / or liver fibrosis in patients with VADS cancer, in order to investigate their impact on the morbidity after treatment of squamous cell carcinomas of the head and neck.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age
* Supported in the department of Orl & CCF or Maxillo-Faciale surgery of the CHU d'Amiens
* Histological diagnosis of epidermoid carcinoma:

  * From the oral cavity
  * From the oropharynx
  * Hypopharynx
  * Larynx
* Any stage of cancer
* Affiliation to a social security scheme

Exclusion Criteria:

* Patient already treated previously for a cancer of the VADS
* Patient referred to in Articles L. 1121-5 to L. 1121-8 and L. 1122-1-2 of the Public Health Code

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-08-20 (Estimated); Primary Completion 2019-06-20 (Estimated); Study Completion 2019-06-20 (Estimated)

PRIMARY OUTCOMES:
Determine the prevalence, by registry data analysis, of cirrhosis in patients with VADS cancer | 1 day
  Determine the prevalence, by registry data analysis, of cirrhosis in patients with VADS cancer

CONTACTS AND LOCATIONS:
Overall Officials: Cyril PAGE, PhD, Principal Investigator — CHU AMIENS PICARDIE
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France